CLINICAL TRIAL: NCT04824248
Title: The Added Value of a Behavioral Weight Reduction Program to Blended Rehabilitation in Patients With Chronic Low Back Pain: A Randomized Clinical Trial
Brief Title: Weight Reduction in CLBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Rotterdam University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Malfliet Anneleen, Prof. Dr. Anneleen Malfiet, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B.U.N. 1432021000411
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Chronic Low-back Pain; Overweight or Obesity
Keywords: chronic low back pain; chronic pain; physiotherapy; physical therapy; weight reduction; pain management
MeSH Terms: conditions — Overweight; Obesity; Chronic Pain; Weight Loss; Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial, including two comparative, balanced online treatment arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental intervention (Experimental): 10 weeks blended therapy delivered using a blended approach. The blended (online and on site) therapy consists of instructive video's, challenges to complete, 1-on-1 sessions with the therapist, online quizzes, online booklets, and online diaries/workbooks. . The experimental group will receive a behavioral weight reduction program combined with pain neuroscience education plus cognition-targeted exercise therapy. The combined therapy will adhere to guidelines for patient-centered care
  Interventions: Behavioral: Pain Neuroscience Education; Behavioral: Cognition-targeted exercise therapy; Behavioral: Behavioral weight reduction program
- Control intervention (Active Comparator): Identically to the experimental intervention, the therapy is provided in a blended format within 10 weeks. Also identical to the experimental intervention, the control intervention will adhere to guidelines for patient-centered care. The control group will receive pain neuroscience education in combination with cognition-targeted exercise therapy alone.
  Interventions: Behavioral: Pain Neuroscience Education; Behavioral: Cognition-targeted exercise therapy

INTERVENTIONS:
Behavioral: Pain Neuroscience Education — Increase pain coping skills and educating the patients that pain is in the brain, and that hypersensitivity of the central nervous system rather than local tissue damage contributes to their symptoms.
  Other Names: Pain Education
Behavioral: Cognition-targeted exercise therapy — Daily (physical) activity and exercise therapy. To confront the patient with movements and activities that are feared, avoided and/or painful using a gradual and cognition-targeted approach.
Behavioral: Behavioral weight reduction program — Changes in diet, behavior and a physical exercise to reach weight loss. It will include a lifestyle approach, incorporating behavioral theories and constructs to assist and facilitate healthy energy balance related behavior.
  Arms: Experimental intervention

SUMMARY:
We will recruit overweight/ obese participants between the age of 18 and 65 with chronic nonspecific low back pain . The participants will be randomly assigned to one of two interventions (each lasting 10 weeks). All interventions will be delivered in a blended format and will be a combination of online education material and face-to-face sessions with a physical therapist. The first group (experimental intervention) will receive a behavioral weight reduction program combined with pain neuroscience education plus cognition-targeted exercise therapy. Participants in the second group (control intervention) will receive pain neuroscience education and cognition-targeted exercise therapy alone. Allocation to the groups will be at random. Participants and assessors will be blinded for group allocation. The primary outcomes is pain intensity. Secondary outcomes include other pain related outcomes, body composition, physical activity, sedentary behavior, dietary intake and function.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (BMI ≥ 25 kg/m2) or obese (BMI ≥ 30 kg/m2) with chronic low back pain
* Non-specific low back pain for at least 3 months' duration
* Currently seeking care for low back pain
* Native Dutch speaker
* Access to internet and computer/tablet/smartphone

Exclusion Criteria:

* Leg pain of 7 or higher (on a maximum of 10) on a numeric rating scale
* Evidence of specific spinal pathology (e.g., hernia, spinal stenosis, spondylolisthesis, infection, spinal fracture or malignancy)
* Evidence of a severe underlying comorbidity (e.g. diabetes, cardiovascular problems, metabolic diseases)
* BMI ≥ 40 kg/m2
* Being pregnant or given birth in the preceding year
* Currently receiving dietary or exercise interventions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Brief Pain inventory (BPI) | Change from baseline to 6 months (T3) after therapy completion
  Questionnaire for assessing clinical pain
Brief Pain inventory (BPI) | Difference between groups at 6 months (T3) after therapy completion
  Questionnaire for assessing clinical pain

SECONDARY OUTCOMES:
Brief Pain inventory (BPI) | Baseline assessment (T0)
  Questionnaire for assessing clinical pain
Brief Pain inventory (BPI) | T1 assessment directly post treatment (i.e. 10 weeks after baseline)
  Questionnaire for assessing clinical pain
Brief Pain inventory (BPI) | T2-assessment 3 months after therapy completion
  Questionnaire for assessing clinical pain
Brief Pain inventory (BPI) | T3-assessment 6 months after therapy completion
  Questionnaire for assessing clinical pain
Central sensitization inventory (CSI) | Baseline Assessment (T0)
  Questionnaire to asses self-reported signs of central sensitization and its overlapping symptoms.
Central sensitization inventory (CSI) | T1-assessment directly post-treatment (i.e. 10 weeks after baseline)
  Questionnaire to asses self-reported signs of central sensitization and its overlapping symptoms.
Central sensitization inventory (CSI) | T2-assessment 3 months after therapy completion
  Questionnaire to asses self-reported signs of central sensitization and its overlapping symptoms.
Central sensitization inventory (CSI) | T3-assessment 6 months after therapy completion
  Questionnaire to asses self-reported signs of central sensitization and its overlapping symptoms.
TANITA Bio-electrical Impedance Analyzer | Baseline assessment (T0)
  Body weight measurement used to calculate BMI (= weight[kg] / height[m]²)
TANITA Bio-electrical Impedance Analyzer | T1-assessment directly post-treatment (i.e. 10 weeks after baseline)
  Body weight measurement used to calculate BMI (= weight[kg] / height[m]²)
TANITA Bio-electrical Impedance Analyzer | T3-assessment 6 months after therapy completion
  Body weight measurement used to calculate BMI (= weight[kg] / height[m]²)
SECA wall-fixed SECA wall-fixed stadiometer | Baseline measurement
  Body height measurement used to calculate BMI (= weight[kg] / height[m]²)
SECA wall-fixed SECA wall-fixed stadiometer | T1-assessment directly post-treatment (i.e. 10 weeks after baseline)
  Body height measurement used to calculate BMI (= weight[kg] / height[m]²)
SECA wall-fixed SECA wall-fixed stadiometer | T3-assessment 6 months after therapy completion
  Body height measurement used to calculate BMI (= weight[kg] / height[m]²)
TANITA MC-780SMA Bio-electrical Impedance Analyzer - body fat | Baseline
  Body composition measurement - body fat
TANITA MC-780SMA Bio-electrical Impedance Analyzer - body fat | T1-assessment directly post-treatment (i.e. 10 weeks after baseline)
  Body composition measurement - body fat
TANITA MC-780SMA Bio-electrical Impedance Analyzer - body fat | T3-assessment 6 months after therapy completion
  Body composition measurement - body fat
TANITA MC-780SMA Bio-electrical Impedance Analyzer - fat free mass | Baseline
  Body composition measurement - fat free mass
TANITA MC-780SMA Bio-electrical Impedance Analyzer - fat free mass | T1-assessment directly post-treatment (i.e. 10 weeks after baseline)
  Body composition measurement - fat free mass
TANITA MC-780SMA Bio-electrical Impedance Analyzer - fat free mass | T3-assessment 6 months after therapy completion
  Body composition measurement - fat free mass
TANITA MC-780SMA Bio-electrical Impedance Analyzer - hydration status | Baseline
  Body composition measurement - hydration status
TANITA MC-780SMA Bio-electrical Impedance Analyzer - hydration status | T1-assessment directly post-treatment (i.e. 10 weeks after baseline)
  Body composition measurement - hydration status
TANITA MC-780SMA Bio-electrical Impedance Analyzer - hydration status | T3-assessment 6 months after therapy completion
  Body composition measurement - hydration status
Food Frequency Questionnaire | Baseline
  Self report questionnaire to asses dietary intake
Food Frequency Questionnaire | T1-assessment directly post-treatment (i.e. 10 weeks after baseline)
  Self report questionnaire to asses dietary intake
Food Frequency Questionnaire | T2-assessment 3 months after therapy completion
  Self report questionnaire to asses dietary intake
Food Frequency Questionnaire | T3-assessment 6 months after therapy completion
  Self report questionnaire to asses dietary intake
International Physical Activity Questionnaire (IPAQ) | Baseline
  Self report questionnaire to asses physical activity
International Physical Activity Questionnaire (IPAQ) | T1-assessment directly post-treatment (i.e. 10 weeks after baseline)
  Self report questionnaire to asses physical activity
International Physical Activity Questionnaire (IPAQ) | T2-assessment 3 months after therapy completion
  Self report questionnaire to asses physical activity
International Physical Activity Questionnaire (IPAQ) | T3-assessment 6 months after therapy completion
  Self report questionnaire to asses physical activity
Sedentary Behavior Questionnaire of Busschaert et a | Baseline
  Self report questionnaire to asses sedentary behavior
Sedentary Behavior Questionnaire of Busschaert et a | T1-assessment directly post-treatment (i.e. 10 weeks after baseline)
  Self report questionnaire to asses sedentary behavior
Sedentary Behavior Questionnaire of Busschaert et a | T2-assessment 3 months after therapy completion
  Self report questionnaire to asses sedentary behavior
Sedentary Behavior Questionnaire of Busschaert et a | T3-assessment 6 months after therapy completion
  Self report questionnaire to asses sedentary behavior
The Short Form Health Survey-36 items (SF-36) | Baseline
  Self report questionnaire to evaluate functional status and well-being or quality of life
The Short Form Health Survey-36 items (SF-36) | T1-assessment directly post-treatment (i.e. 10 weeks after baseline)
  Self report questionnaire to evaluate functional status and well-being or quality of life
The Short Form Health Survey-36 items (SF-36) | T2-assessment 3 months after therapy completion
  Self report questionnaire to evaluate functional status and well-being or quality of life
The Short Form Health Survey-36 items (SF-36) | T3-assessment 6 months after therapy completion
  Self report questionnaire to evaluate functional status and well-being or quality of life
Fear avoidance Beliefs Questionnaire | Baseline
  Self report questionnaire to evaluate fear avoidance beliefs. Total score: 0 - 96 (min-max) Work Subscore: 0 - 66 (min-max) Physical Activity Subscore: 0 - 30 (min-max) Higher scores indicate more fear, pain and disability.
Fear avoidance Beliefs Questionnaire | T1-assessment directly post-treatment (i.e. 10 weeks after baseline)
  Self report questionnaire to evaluate fear avoidance beliefs. Total score: 0 - 96 (min-max) Work Subscore: 0 - 66 (min-max) Physical Activity Subscore: 0 - 30 (min-max) Higher scores indicate more fear, pain and disability.
Fear avoidance Beliefs Questionnaire | T2-assessment 3 months after therapy completion
  Self report questionnaire to evaluate fear avoidance beliefs. Total score: 0 - 96 (min-max) Work Subscore: 0 - 66 (min-max) Physical Activity Subscore: 0 - 30 (min-max) Higher scores indicate more fear, pain and disability.
Fear avoidance Beliefs Questionnaire | T3-assessment 6 months after therapy completion
  Self report questionnaire to evaluate fear avoidance beliefs. Total score: 0 - 96 (min-max) Work Subscore: 0 - 66 (min-max) Physical Activity Subscore: 0 - 30 (min-max) Higher scores indicate more fear, pain and disability.

CONTACTS AND LOCATIONS:
Locations (2):
- Vrije Universiteit Brussel, Brussels, Belgium
- Rotterdam University of Applied Sciences, Rotterdam, Netherlands